CLINICAL TRIAL: NCT04789720
Title: Using Information Technology to Improve Outcomes for Children Living With Cancer
Acronym: SyMon-SAYS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Ann & Robert H Lurie Children's Hospital of Chicago (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jin-Shei Lai, Profesor, Medical Social Sciences and Pediatrics, Northwestern University Feinberg School of Medicine., Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1U01CA246612-01 (NIH); 1U01CA246612-01 (NIH)
Record Dates: First submitted 2021-02-05; First posted 2021-03-10 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Cancer
Keywords: children living with cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to Group A (SyMon-SAYS intervention) or B (waitlist-control), stratified by gender, age (8-12 vs 13-17), and type of cancer (brain tumor vs. leukemia vs. others). To achieve allocation concealment, the computer-based data management system will assign participants to one of two groups after the study enrollment procedures. A permuted block sequence will be used. Participants will be informed of their group assignment (Group A or B) after the baseline assessment. Participants will complete a 9-item SyMon-SAYS Weekly Symptom Assessment Scale via Epic MyChart patient portal during the intervention phase (Group A: Wk1-16 or Group B: Wk9-16)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SyMon-SAYS Intervention (Group A) (Experimental): Group A participants will receive the SyMon-SAYS intervention every week for 16 weeks.
  Interventions: Behavioral: Symptom Monitoring & Systematic Assessment and Reporting System in Young Survivors (SyMon-SAYS)
- SyMon-SAYS Waitlist Control (Group B) (Other): The waitlist control group participants (Group B) will receive their usual care during weeks 1-8 and will receive the SyMon-SAYS intervention every week during weeks 9-16.
  Interventions: Behavioral: Symptom Monitoring & Systematic Assessment and Reporting System in Young Survivors (SyMon-SAYS)

INTERVENTIONS:
Behavioral: Symptom Monitoring & Systematic Assessment and Reporting System in Young Survivors (SyMon-SAYS) — Participants will complete a 9-item SyMon-SAYS symptom assessment checklist every week during the intervention phase (Intervention Group: weeks 1-16; Waitlist Control: weeks 9-16) through Epic MyChart via mobile app, computer or tablet. Patients' symptom scores will be monitored and reported to their oncology care providers. When a patient symptom score trigger threshold is met, the system will generate an email alert through Epic (electronic medical record system) messaging to the provider. The provider will take appropriate actions using his/her clinical judgement, including contacting patients and families when needed. Symptom scores overtime will be available in MyChart (patient-facing component of the Epic electronic medical record system) for patients and parents to review and to discuss with the child's provider during clinical visits.

SUMMARY:
This proposed study plans to develop and evaluate a patient-oriented, technology-based, symptom monitoring system that reports symptoms experienced by children with cancer to their parents and health care providers.

DETAILED DESCRIPTION:
Cancer is a leading cause of death and disability in children under 15 years of age. Its unrelieved symptoms and side effects of often-aggressive treatments can lead to poor psychosocial functioning and decreased health-related quality of life (HRQOL) for patients and their families. Barriers at the patient, healthcare provider and system levels can contribute to poor symptom management. A technology-based program can minimize these barriers by routinely collecting and interpreting patient-reported outcomes (PROs) and patient/parent contextual data in pediatric oncology ambulatory settings in a manner that is efficient, actionable by physicians, supports engagement of patients and families with their health and care, and improves clinical processes and outcomes. This proposed project will develop and evaluate the effectiveness of such a program: Symptom Monitoring & Systematic Assessment and Reporting System in Young Survivors (SyMon-SAYS). We hypothesize that the SyMon-SAYS intervention will decrease parent-perceived barriers to managing their child's symptoms, decrease patient symptom burden, increase patients' and parents' self-efficacy, and ultimately increase patient HRQOL.

ELIGIBILITY:
Inclusion Criteria:

Patients

* Have an hematology/oncologic diagnosis (including a brain tumor)
* Be on-treatment or within 6 months post-therapy
* Be between 8 and 17 years old
* English-speaking
* Have sufficient cognitive and motor abilities to complete survey via an electronic device (e.g., smartphone, iPAD, etc.) or computer
* Be able and willing to sign assent forms (for those 12-17 years old).

Parent/legal guardian

* Be a parent (father or mother) or a legal guardian of eligible patients
* Demonstrates sufficient English and/or Spanish ability to understand and sign the informed consent form
* Have sufficient cognitive and motor abilities to complete survey via an electronic device (e.g., smartphone, iPAD, etc) or computer

Exclusion Criteria:

* Patients who cannot understand English sufficiently to sign consent/assent form
* Patients who cannot understand English sufficiently to complete the questionnaires

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 216 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Adherence to intervention | 16 weeks for Group A and 8 weeks for Group B
  The adherence to the SyMon-SAYS Intervention will be evaluated by using the percentage of dyads completing the symptom assessments at all time-points (16 weeks for Group A participants and 8 weeks for Group B participants), excluding those who are off-study or deceased.
Overall symptom burden | change from baseline to week 8; and from week 9 to week 16
  Evidence of decreased or maintained symptom burden as measured by the SyMon-SAYS symptom checklist from baseline to week 8 (primary analysis) and from week 9 to week 16. Each symptom is rated by using a 5-point rating scale and will be evaluated separately. Higher scores represent worse symptom burden.
Perceived symptom management barriers as reported by parents of patients | change from baseline to week 8; and from week 9 to week 16
  Evidence of decreased or maintained perceived symptom barriers as measured by a modified 23-item Symptom Management Barriers Questionnaire checklist from baseline to week 8 (primary analysis) and from week 9 to week 19. Possible scores range from 23 - 115. Higher scores represent more perceived barriers.
Health related quality of life | change from baseline to week 8; and from week 9 to week 16
  Evidence of improved or maintained health related quality of life (physical function, fatigue, depressive symptom, anxiety, anger, social functioning), as measured by the pediatric Patient Reported Outcome Measurement Information System, PROMIS, (child self-report version) from baseline to week 8 as well as from week 9 to week 16. Scores will be reported by using a T-score system, in which mean of the norming group =50 and SD=10. Higher scores represent better functioning (mobility, upper extremity function, peer relationships) or worse symptoms (depression, anxiety, anger and fatigue).
Self-Efficacy | change from baseline to week 8; and from week 9 to week 16
  Evidence of improved or maintained self-efficacy in managing symptoms related to cancer therapy as measured by using the NIH Toolbox Self-Efficacy (child self-reported version) from baseline to week 8 and from week 9 to week 16. Scores will be reported by using a T-score metric, with a general population mean=50 and SD=10. Higher scores represent better self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Shei Lai, PhD, Principal Investigator — Northwestern University
Locations (1):
- Ann & Robert H. Lurie Childrens Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lai JS, Jensen SE, Peipert JD, Mitchell SA, Garcia SF, Cella D, Goldman S, Lenzen A. Using IT to Improve Outcomes for Children Living With Cancer (SyMon-SAYS): Protocol for a Single-Institution Waitlist Randomized Controlled Trial. JMIR Res Protoc. 2023 Sep 8;12:e50993. doi: 10.2196/50993. PMID 37682593

DOCUMENTS (2):
  • Informed Consent Form: Parental Consent (2024-09-09): https://cdn.clinicaltrials.gov/large-docs/20/NCT04789720/ICF_002.pdf
  • Informed Consent Form: Adolescent Assent (2024-09-09): https://cdn.clinicaltrials.gov/large-docs/20/NCT04789720/ICF_003.pdf